CLINICAL TRIAL: NCT04314648
Title: Pilot Test of a Substance Use Treatment and Recovery Team (START) for Medical Inpatients With Opioid and Alcohol Use Disorders
Brief Title: Substance Use Treatment and Recovery Team (START)
Acronym: START
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Cedars-Sinai Medical Center (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCAAD013; 1R34DA047492-01 (NIH)
Record Dates: First submitted 2020-03-16; First posted 2020-03-19 (Actual); Results first posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-03

CONDITIONS: Opioid-use Disorder; Opioid-Related Disorders; Alcohol Use Disorder; Alcohol-Related Disorders
Keywords: Collaborative Care; Hospital; Addiction; Opioid Use Disorder; Alcohol Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders; Alcoholism; Alcohol-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- START (Active Comparator): START is a model of care based on Collaborative Care. START is team driven, population-focused, measurement based, and focused on promoting adoption of evidence-based interventions. The purpose of this model is to increase adoption of evidence-based interventions for opioid and alcohol use disorders, and to increase linkage to aftercare.
  The components of the START intervention are as follows:
  1. Triage
  2. Engage, Assess, and Plan
  3. Treat
  4. Communicate and Coordinate
  5. Follow up
  6. Monitor
  Interventions: Behavioral: Substance Use Treatment and Recovery Team (START)
- Usual Care (No Intervention): Usual care for people with alcohol or opioid use disorder.

INTERVENTIONS:
Behavioral: Substance Use Treatment and Recovery Team (START) — Embedding of a collaborative care team, called the Substance Use Treatment and Recovery Team (START), for inpatients with OAUDs within an existing hospital consultation liaison psychiatry service.
  Arms: START

SUMMARY:
Despite high prevalence, few hospitalized inpatients with opioid or alcohol use disorders (OAUDs) receive evidence-based treatments while in the hospital or get linked with appropriate follow-up care, leading to poor clinical outcomes and high readmission rates and costs. The purpose of this study is to evaluate whether a physician and care manager with addiction expertise, both members of the Substance Abuse Treatment and Recovery Team (START), can help improve initiation of treatment in the hospital and linkage to follow-up care upon discharge. START members have expertise in the treatment of substance use disorders.

START will work with the medical or surgical team to ensure appropriate care is received. That care will include therapy, focused discharge planning, and medication treatment options. START will also help establish a follow-up plan for continuation of treatment after hospital discharge.

To assess feasibility, the study will enroll 80 patients admitted to the hospital over 5 months in a pilot randomized clinical trial and collect baseline and 1-month follow-up data. To determine acceptability, the study will conduct semi-structured interviews with 40 providers. Results of this pilot study will inform a larger clinical trial.

DETAILED DESCRIPTION:
The specific aims of this three-year R34 are to prepare for a clinical trial by (1) developing the protocol and resources for Substance Use Treatment and Recovery Team (START) to address untreated opioid or alcohol use disorders (OAUDs) among hospitalized inpatients and actively link them to follow-up care, and by (2) conducting a pilot RCT to assess (a) implementation feasibility; and (b) acceptability among patients and providers. The study is of critical importance to public health because millions of people in the United States need, but do not receive, treatment for substance-use disorders. OAUDs are of particular concern because of high rates of morbidity, mortality, hospitalizations, and readmissions, as well as the increasing incidence of opioid-use disorders and associated medical consequences and overdose deaths. Moreover, OAUDs are common substance use disorders among medical inpatients.

However, despite high prevalence, few inpatients with OAUDs receive evidence-based treatments while in the hospital. Most physicians and other providers in acute hospital settings are not trained to assess or manage patients with OAUDs, contributing to low rates of OAUD identification and treatment initiation. Pharmacotherapies to address OAUDs are effective for use across medical settings but are seldom initiated in hospitals or recommended as part of follow-up care. Inpatient hospitalization offers a pivotal opportunity to decrease unmet need. Starting treatment in the hospital and effectively linking patients with follow-up care could not only improve outcomes, but also could decrease high rates of hospital readmission and ultimately lower costs.

The current standard of care for hospitalized patients with OAUD-screening, brief intervention and referral to treatment-is not effective for those with OAUDs, possibly because it does not include initiation of medication or facilitate linkage to follow-up OAUD care. Barriers to OAUD treatment for inpatients may include lack of expertise on the medical team, absence of an organized system for assessing and treating patients with OAUD, patient ambivalence about treatment, and lack of follow-up after discharge. The START will consist of an physician and care manager team with OAUD expertise who provide population-focused monitoring and measurement-based decision-making to support the medical team.

START will use evidence-based components, including a motivational interviewing-based therapeutic intervention, targeted discharge planning, and active referral.

To develop the protocol, we will draw from our prior work in primary care and other evidence-based resources, and obtain input from a stakeholder advisory board comprised of patients and providers. To assess feasibility, we will enroll 80 patients admitted to the hospital over 5 months in a pilot RCT and collect baseline and 1-month follow-up data.

To determine acceptability, we will conduct interviews with providers and patients. The proposed study would be the first to test a consultation-liaison service-based START to improve care for inpatients with OAUD.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient at CSMC
* Age 18 and older
* Screens positive for moderate to severe OAUDs based on the alcohol and opioid questions on the
* World Health Organization (WHO) Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST).
* Speaks English as primary language
* The usual attending physician agrees to patient's participation
* Has decision-making capacity and is not gravely disabled

Exclusion Criteria:

* Currently receiving FDA-approved medication treatment for an opioid or alcohol use disorder
* Gravely disabled (per clinical judgement)
* Does not have decision-making capacity (per clinical judgement)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison J Ober, PhD, Principal Investigator — RAND; Itai Danovitch, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make the data and associated documentation available to users under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying the data after analyses are completed.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be available upon completion of analyses until five years after study completion.
Access Criteria: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying the data after analyses are completed.

RESULTS

PARTICIPANT FLOW:
Groups:
- START: START is a model of care based on Collaborative Care. START is team driven, population-focused, measurement based, and focused on promoting adoption of evidence-based interventions. The purpose of this model is to increase adoption of evidence-based interventions for opioid and alcohol use disorders, and to increase linkage to aftercare.
  The components of the START intervention are as follows:
  1. Triage
  2. Engage, Assess, and Plan
  3. Treat
  4. Communicate and Coordinate
  5. Follow up
  6. Monitor
  Substance Use Treatment and Recovery Team (START): Embedding of a collaborative care team, called the Substance Use Treatment and Recovery Team (START), for inpatients with OAUDs within an existing hospital consultation liaison psychiatry service.
Period: Overall Study
Arm/Group | START | Usual Care
Started | 38 | 50
Completed | 38 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | START | Usual Care | Total
Number analyzed (Participants) | 38 | 50 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (12.9) | 44.5 (13.2) | 44.5 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 26 | 40 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 18 | 28
  Not Hispanic or Latino | 28 | 32 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 31 | 43 | 74
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 38 | 50 | 88
Heavy Drinking among Patients with Alcohol Use Disorder [Count of Participants; unit: Participants] — For men, consuming an average of more than two drinks per day; for women, consuming an average of more than one drink per day during the reporting period of 30 days, extended from the NIAAA definition of this level of drinking over 14 days) (National Institute on Alcohol Abuse and Alcoholism, 2022). Obtained by combining the separate survey questions of # of days drinking and # of drinks per day in past 30 days) (binary) Population: Number analyzed is patients with an alcohol use disorder (minus one patient who did not respond to this question)
  Participants
    number analyzed (Participants) | 31 | 41 | 72
    (all) | 26 | 32 | 58
Any Days of Opioid Use among Patients with Opioid Use Disorder [Count of Participants; unit: Participants] — Population: Number analyzed is patients with opioid use disorder.
  Participants
    number analyzed (Participants) | 13 | 14 | 27
    (all) | 9 | 11 | 20
Days of Alcohol Use among Patients with Alcohol Use Disorder [Mean (Standard Deviation); unit: Days of Use] — Population: Number analyzed is patients with an alcohol use disorder.
  Days of Use
    number analyzed (Participants) | 31 | 42 | 73
    (all) | 18.39 (10.34) | 21.21 (10.65) | 20.01 (10.54)
Number of Drinks per Day among those with Alcohol Use Disorder who Drank in the Past 30 Days [Mean (Standard Deviation); unit: Drinks per Day] — Population: Number analyzed is patients with an alcohol use disorder
  Drinks per Day
    number analyzed (Participants) | 28 | 38 | 66
    (all) | 10.21 (7.33) | 9.97 (7.70) | 10.08 (7.49)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With In-hospital Initiation of Medication for OUD or AUD
Description: Received medication for an OUD or AUD between admission and discharge (Binary)
Time Frame: During the inpatient stay, an average of 7 days
Population: All study participants.
Measure: Count of Participants; unit: Participants
Arm/Group | START | Usual Care
Number analyzed (Participants) | 38 | 50
Participants | 22 | 9
Statistical Analysis 1: Comparison: START vs Usual Care; Test type: Superiority; p < .001, Regression, Logistic; Odds Ratio (OR) = 6.26, 95% CI 2-sided [2.38 to 16.48]

2. Primary Outcome: Number of Patients With Linkage to Follow-up Care for OUD or AUD
Description: Received at least one visit post-discharge for medication and/or psychosocial care for OUD or AUD (Binary)
Time Frame: 30 days post-discharge
Population: Study participants who received a 1-month follow-up interview.
Measure: Count of Participants; unit: Participants
Arm/Group | START | Usual Care
Number analyzed (Participants) | 29 | 44
Participants | 24 | 20
Statistical Analysis 1: Comparison: START vs Usual Care; Test type: Superiority; p < .01, Regression, Logistic; Odds Ratio, log = 5.76, 95% CI 2-sided [1.86 to 17.86]

3. Primary Outcome: Number of Patients With Heavy Drinking in Past 30-days at Follow-up Among Patients With Alcohol Use Disorder
Description: For men, consuming an average of more than two drinks per day; for women, consuming an average of more than one drink per day during the reporting period of 30 days, extended from the NIAAA definition of this level of drinking over 14 days), among patients with alcohol use disorder at follow-up (National Institute on Alcohol Abuse and Alcoholism, 2022). Obtained by combining the separate survey questions of # of days drinking and # of drinks per day in past 30 days) (binary)
Time Frame: 30-days post-discharge
Population: Study participants with an alcohol use disorder who received a 1-month follow-up interview.
Measure: Count of Participants; unit: Participants
Arm/Group | START | Usual Care
Number analyzed (Participants) | 24 | 36
Participants | 5 | 9
Statistical Analysis 1: Comparison: START vs Usual Care; Test type: Superiority; p = .64, Regression, Logistic; Odds Ratio (OR) = .74, 95% CI 2-sided [.21 to 2.64] — Main effects of the intervention on this outcome were compared between arms by fitting follow-up values to a logistic regression model, adjusted for baseline use

4. Primary Outcome: Number of Patients With Any Days of Opioid Use in Past 30-days at Follow-up Among Patients With Opioid Use Disorder
Description: Any days using opioids at follow-up, based on NSDUH 30-day substance use questions (Center for Behavioral Health Statistics and Quality, 2018), (binary)
Time Frame: 30 days post-discharge
Population: Study participants with opioid use disorder who received a 1-month follow-up interview.
Measure: Count of Participants; unit: Participants
Arm/Group | START | Usual Care
Number analyzed (Participants) | 11 | 12
Participants | 5 | 5
Statistical Analysis 1: Comparison: START vs Usual Care; Test type: Superiority; p = .35, Regression, Logistic; Odds Ratio (OR) = 2.67, 95% CI 2-sided [.35 to 20.51] — [estimate comment as in outcome 3, analysis 1]

5. Primary Outcome: Average Number of Days of Alcohol Use in Past 30-Days at Follow-Up Among Patients With Alcohol Use Disorder
Description: Number of days of any alcohol use in the past 30 days at follow-up among patients with an alcohol use disorder
Time Frame: 30-days post-discharge
Population: Study participants with alcohol use disorder who received a 1-month follow-up interview.
Measure: Mean (Standard Deviation); unit: Days of use
Arm/Group | START | Usual Care
Number analyzed (Participants) | 24 | 37
Days of use | 4.08 (7.57) | 6.24 (9.37)
Statistical Analysis 1: Comparison: START vs Usual Care; Test type: Superiority; p = .43, Regression, Linear; Mean Difference (Net) = -1.85, Standard Error of Mean 2.32 — Main effects of the intervention on this outcome were compared between arms by fitting follow-up values to a linear regression model, adjusted for baseline use

6. Primary Outcome: Average Number of Drinks Per Day in Past 30-days at Follow-up Among Patients With Alcohol Use Disorder
Description: Number of drinks per day among those with alcohol use disorder who drank in the past 30 days at follow-up
Time Frame: 30-days post-discharge
Population: Study participants with alcohol use disorder who drank in the past 30 days and received a 1-month follow-up interview.
Measure: Mean (Standard Deviation); unit: Drinks per day
Arm/Group | START | Usual Care
Number analyzed (Participants) | 11 | 17
Drinks per day | 9.82 (9.60) | 7.00 (7.16)
Statistical Analysis 1: Comparison: START vs Usual Care; Test type: Superiority; p = .44, Regression, Linear; Mean Difference (Net) = 2.35, Standard Error of Mean 3.00 — Main effects of the intervention on this outcome were compared between arms by fitting follow-up values to a liner regression model, adjusted for baseline use

7. Secondary Outcome: Number of Patients Readmitted to Cedars-Sinai Medical Center (CSMC) Within 90 Days After Discharge
Description: Patient was readmitted to Cedars Sinai Medical Center (the same hospital) for any reason, up to 90-days after discharge
Time Frame: 90 days post-discharge
Population: All study participants.
Measure: Count of Participants; unit: Participants
Arm/Group | START | Usual Care
Number analyzed (Participants) | 38 | 50
Participants | 7 | 8
Statistical Analysis 1: Comparison: START vs Usual Care; Test type: Superiority; p = .77, Regression, Logistic; Odds Ratio (OR) = 1.19, 95% CI 2-sided [.39 to 3.62]

ADVERSE EVENTS:
Time Frame: Ten months
Arm/Group | START | Usual Care
All-Cause Mortality (participants affected / at risk) | 2/38 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/50
Other Adverse Events (participants affected / at risk) | 0/38 | 0/50

LIMITATIONS AND CAVEATS:
The pilot sample size is small and combines individuals with AUD and OUD. The follow-up period was only one month after hospital discharge. Readmission was measured at only the admitting hospital. While the ASSIST, used to assess OUD and AUD, has been validated in the primary care setting, it has not be validated in the hospital setting. Use of the NSDUH 30-day use questions to measure self-reported opioid and alcohol use may have resulted in underreporting at both baseline and follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/48/NCT04314648/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-27): https://cdn.clinicaltrials.gov/large-docs/48/NCT04314648/ICF_001.pdf